CLINICAL TRIAL: NCT02784704
Title: A Phase 3, Randomized, Double-Blind, Double-Dummy, Multicenter, Prospective Study to Assess the Efficacy and Safety of Eravacycline Compared With Meropenem in Complicated Intra-abdominal Infections
Brief Title: Efficacy and Safety Study of Eravacycline Compared With Meropenem in Complicated Intra-abdominal Infections
Acronym: IGNITE4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tetraphase Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Organization: La Jolla Pharmaceutical Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP-434-025
Record Dates: First submitted 2016-05-23; First posted 2016-05-27 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Complicated Intra-abdominal Infections; Complicated Appendicitis
MeSH Terms: interventions — eravacycline; Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eravacycline (Experimental)
  Interventions: Drug: Eravacycline; Drug: Placebo
- Meropenem (Active Comparator)
  Interventions: Drug: Meropenem; Drug: Placebo

INTERVENTIONS:
Drug: Eravacycline
  Other Names: TP-434
  Arms: Eravacycline
Drug: Meropenem
  Other Names: Merrem
  Arms: Meropenem
Drug: Placebo

SUMMARY:
This is a Phase 3, randomized, double-blind, double-dummy, multicenter, prospective study to assess the efficacy, safety, and pharmacokinetics (PK) of eravacycline compared with meropenem in the treatment of complicated intra-abdominal infections (cIAIs).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant hospitalized for cIAI
* At least 18 years of age
* Evidence of a systemic inflammatory response
* Abdominal pain or flank pain (with or without rebound tenderness), or pain caused by cIAI that is referred to another anatomic area
* Able to provide informed consent
* If male: must agree to use an effective barrier method of contraception during the study and for 14 days following the last dose if sexually active with a female of childbearing potential
* If female, not pregnant or nursing or, if of childbearing potential: either will commit to use at least two medically accepted, effective methods of birth control (for example, condom, oral contraceptive, indwelling intrauterine device, hormonal implant /patch, injections, approved cervical ring) during study drug dosing and for 14 days following last study drug dose or practicing sexual abstinence

Exclusion Criteria:

* Unlikely to survive the 6-8 week study period
* Creatinine clearance of ≤50 milliliter (mL)/minute
* Presence or possible signs of significant hepatic disease
* Immunocompromised condition, including known human immunodeficiency virus (HIV) positivity, transplant recipients, and hematological malignancy
* History of moderate or severe hypersensitivity reactions to tetracyclines, carbapenems, β-lactam antibiotics, or to any of the excipients contained in the study drug formulations
* Participation in any investigational drug or device study within 30 days prior to study entry
* Known or suspected current central nervous system (CNS) disorder that may predispose to seizures or lower seizure threshold (for example, severe cerebral arteriosclerosis, epilepsy)
* Antibiotic-related exclusions:

  1. Receipt of effective antibacterial drug therapy for cIAI for a continuous duration of >24-hours during the 72-hours preceding randomization [however, participants with documented cIAI (that is, known baseline pathogen) who have received at least 72-hours of antibiotic therapy and are considered treatment failures may be enrolled. Treatment failure is defined as persistent fever and/or clinical symptoms; or the development of a new intra-abdominal abscess after ≥72-hours of antibiotic therapy], or
  2. Receipt of meropenem or any other carbapenem, or tigecycline for the current infection, or
  3. Need for concomitant systemic antimicrobial agents effective in cIAI other than study drug
* Refusal of mechanical ventilation, dialysis or hemofiltration, cardioversion, or any other resuscitative measures and drug/fluid therapy at time of consent
* Known or suspected inflammatory bowel disease or associated visceral abscess
* The anticipated need for systemic antibiotics for a duration of more than 14 days
* Systemic malignancy that required chemotherapy, immunotherapy, radiation therapy, or antineoplastic therapy within the previous 3 months or that is anticipated to begin prior to the Test-of-Cure (TOC) visit
* Known at study entry to have cIAI caused by a pathogen(s) resistant to one of the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2017-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Tetraphase Pharmaceuticals
Locations (54):
- United States (6):
  - Los Angeles, California
  - Indianapolis, Indiana
  - Las Vegas, Nevada
  - Somers Point, New Jersey
  - Cleveland, Ohio
  - Columbus, Ohio
- Bulgaria (5):
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
  - Varna
- Czechia (4):
  - Jihlava
  - Kladno
  - Kolín
  - Prague
- Estonia (4):
  - Tallinn
  - Tartu
  - Viljandi
  - Võru
- Georgia (4):
  - Batumi
  - Kutaisi
  - Tbilisi
  - Zugdidi
- Hungary (4):
  - Győr
  - Kaposvár
  - Pécs
  - Veszprém
- Latvia (4):
  - Daugavpils
  - Liepāja
  - Rēzekne
  - Riga
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Romania (5):
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Târgu Mureş
  - Timișoara
- Russia (7):
  - Arkhangelsk
  - Kaluga
  - Krasnodar
  - Nizhny Novgorod
  - Saint Petersburg
  - Volgograd
  - Vsevolozhsk
- Ukraine (8):
  - Dnipro
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
  - Lviv
  - Odesa
  - Uzhhorod
  - Vinnytsia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Solomkin JS, Gardovskis J, Lawrence K, Montravers P, Sway A, Evans D, Tsai L. IGNITE4: Results of a Phase 3, Randomized, Multicenter, Prospective Trial of Eravacycline vs Meropenem in the Treatment of Complicated Intraabdominal Infections. Clin Infect Dis. 2019 Aug 30;69(6):921-929. doi: 10.1093/cid/ciy1029. PMID 30561562
- [Derived] Solomkin JS, Sway A, Lawrence K, Olesky M, Izmailyan S, Tsai L. Eravacycline: a new treatment option for complicated intra-abdominal infections in the age of multidrug resistance. Future Microbiol. 2019 Oct;14:1293-1308. doi: 10.2217/fmb-2019-0135. Epub 2019 Oct 1. PMID 31570004
- See also: IGNITE4: Results of a Phase 3, Randomized, Multicenter, Prospective Trial of Eravacycline vs. Meropenem in the Treatment of Complicated Intra-Abdominal Infections — https://www.ncbi.nlm.nih.gov/pubmed/?term=30561562

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with a diagnosis of complicated intra-abdominal infection (cIAI) requiring surgery were recruited into this study. Subjects were recruited in 65 centers worldwide. The first subject enrolled on 13 October 2016 and the last subject completed on 19 May 2017.
Groups:
- Eravacycline: Eravacycline 1.0mg/kg q12h
- Meropenem: Meropenem 1g q8h
Period: Overall Study
Arm/Group | Eravacycline | Meropenem
Started | 250 | 250
Treated | 250 | 249
Completed | 237 | 241
Not Completed | 13 | 9
Not completed — Adverse Event | 4 | 2
Not completed — Lost to Follow-up | 6 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Subject Non Compliance | 2 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat Population: all randomized subjects who receive any amount of study drug.
Groups:
- Eravacycline: Eravacycline 1.0 mg/kg q12h
- Meropenem: Meropenem 1 g q8h
- Total: Total of all reporting groups
Arm/Group | Eravacycline | Meropenem | Total
Number analyzed (Participants) | 250 | 249 | 499
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 180 | 174 | 354
  >=65 years | 70 | 75 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (17.69) | 52.8 (18.24) | 52.4 (17.931)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 120 | 231
  Male | 139 | 129 | 268
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 239 | 238 | 477
  Unknown or Not Reported | 7 | 11 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 249 | 249 | 498
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Latvia | 34 | 33 | 67
  Romania | 23 | 34 | 57
  Hungary | 10 | 20 | 30
  United States | 8 | 4 | 12
  Czechia | 13 | 16 | 29
  Ukraine | 39 | 43 | 82
  Georgia | 8 | 16 | 24
  Bulgaria | 52 | 41 | 93
  Lithuania | 22 | 18 | 40
  Estonia | 20 | 11 | 31
  Russia | 21 | 13 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Favorable Clinical Response at the Test-of-Cure (TOC) Visit in the Microbiological Intent-to-treat (Micro-ITT) Population
Description: Clinical cure was defined as complete resolution or significant improvement of signs and symptoms of the index infection such that no additional antibacterial therapy, surgical, or radiological intervention was required.
  Clinical failure was defined as death related to complicated intra-abdominal infection (cIAI), persistence of clinical symptoms of cIAI, unplanned surgical or percutaneous drainage procedures for complication or recurrence of cIAI, post-surgical wound infections requiring systemic antibiotics, or initiation of rescue antibacterial drug therapy for treatment of cIAI.
  Indeterminate/missing was defined as an outcome that was neither a clinical cure nor clinical failure, if the investigator did not complete an assessment, if a study visit was not conducted, or if the subject died for a cause unrelated to cIAI.
Time Frame: TOC visit: 25-31 days after first dose of study drug
Population: Microbiological Intent-to-Treat Population: all randomized subjects who have at least one baseline bacterial pathogen that causes cIAI and against which the investigational drug has in vitro antibacterial activity.
Measure: Count of Participants; unit: Participants
Arm/Group | Eravacycline | Meropenem
Number analyzed (Participants) | 195 | 205
Participants
  Clinical Cure | 177 | 187
  Clinical Failure | 7 | 7
  Indeterminate/missing | 11 | 11

2. Secondary Outcome: Number of Participants With a Favorable Clinical Response at the Test-of-Cure (TOC) Visit in the All-Treated (MITT) Population
Description: as for outcome 1
Time Frame: TOC visit: 25-31 days after first dose of study drug
Population: Modified Intent-to-Treat Population: all randomized subjects who receive any amount of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Meropenem: Meropenem 1.0g q8h
Arm/Group | Eravacycline | Meropenem
Number analyzed (Participants) | 250 | 249
Participants
  Clinical Cure | 231 | 228
  Clinical Failure | 7 | 9
  Indeterminate/missing | 12 | 12

3. Secondary Outcome: Number of Participants With a Favorable Clinical Response at the Test-of-Cure (TOC) Visit in the Clinically Evaluable (CE) Population
Description: Clinical cure was defined as complete resolution or significant improvement of signs and symptoms of the index infection such that no additional antibacterial therapy, surgical, or radiological intervention was required.
  Clinical failure was defined as death related to complicated intra-abdominal infection (cIAI), persistence of clinical symptoms of cIAI, unplanned surgical or percutaneous drainage procedures for complication or recurrence of cIAI, post-surgical wound infections requiring systemic antibiotics, or initiation of rescue antibacterial drug therapy for treatment of cIAI.
Time Frame: TOC visit: 25-31 days after first dose of study drug
Population: Clinically Evaluable: all randomized subjects who meet key inclusion/exclusion criteria and follow other important components of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Eravacycline | Meropenem
Number analyzed (Participants) | 225 | 231
Participants
  Clinical Cure | 218 | 222
  Clinical Failure | 7 | 9

ADVERSE EVENTS:
Time Frame: 52 days
Description: All serious adverse events by preferred term, Safety Population
Groups:
- Eravacycline: Eravacycline 1 mg/kg q12h
Arm/Group | Eravacycline | Meropenem
All-Cause Mortality (participants affected / at risk) | 4/250 | 1/249
Serious Adverse Events (participants affected / at risk) | 15/250 | 16/249
Other Adverse Events (participants affected / at risk) | 29/250 | 8/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eravacycline (N=250) | Meropenem (N=249)
Pneumonia (Infections and infestations) | 2 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Neuroendocrine tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Ureteric rupture (Renal and urinary disorders) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal fistula (Gastrointestinal disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Splenic hematoma (Blood and lymphatic system disorders) | 0 | 1
Pelvic fluid collection (Reproductive system and breast disorders) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Suture related complication (Injury, poisoning and procedural complications) | 0 | 1
Wound decomposition (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eravacycline (N=250) | Meropenem (N=249)
Nausea (Gastrointestinal disorders) | 12 | 2
Vomiting (Gastrointestinal disorders) | 9 | 5
Infusion site phlebitis (General disorders) | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications should include input from the PI, his/her colleagues, other PIs in the trial and the Sponsor's personnel; such input should be reflected in the authorship. Agreement of order of authors should be established before writing a manuscript. The PI interested in participating in writing the manuscript should contact the Sponsor. The PI shall not make any publication without the Sponsor's prior written approval, which may be withheld or granted by the Sponsor, in it's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT02784704/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT02784704/SAP_001.pdf